CLINICAL TRIAL: NCT00238342
Title: Pelvic Mass Study to Develop Serum Proteomic Profiles (SIGNATURES) for Epithelial Ovarian Cancer Diagnosis and Prognosis
Brief Title: Proteomic Profiling in Diagnosing Ovarian Cancer in Patients Who Are Undergoing Surgery for an Abnormal Pelvic Mass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000445437; GOG-0220
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2007-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian serous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization; Biopsy

INTERVENTIONS:
Genetic: proteomic profiling
Other: surface-enhanced laser desorption/ionization-time of flight mass spectrometry
Procedure: biopsy

SUMMARY:
RATIONALE: Finding specific proteins in the blood may help doctors tell whether a patient has ovarian cancer.

PURPOSE: This clinical trial is studying how well proteomic profiling works in diagnosing ovarian cancer in patients who are undergoing surgery for an abnormal pelvic mass.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Generate and validate a serum proteomic profile that can predict the presence of invasive ovarian epithelial cancer using preoperative serum specimens obtained from patients undergoing surgical evaluation for an abnormal pelvic mass.

Secondary

* Generate a proteomic profile that can distinguish early- from late-stage invasive ovarian epithelial cancer using preoperative serum specimens from patients who are subsequently diagnosed with invasive ovarian epithelial cancer.

Tertiary

* Determine whether serum proteomic profiling can predict the presence of postoperative residual disease in these patients.
* Determine whether serum proteomic profiling can predict prognosis in these patients.

OUTLINE: This is a pilot, two-part, multicenter study.

* Part A: Within 3 weeks prior to surgical evaluation, patients undergo collection of serum specimen for proteomic profiling using surface-enhanced or matrix-associated laser desorption ionization spectrometry-time of flight detection (SELDI/MALDI-TOF). Patients then undergo surgical evaluation (i.e., biopsy and/or resection) of the pelvic mass. Patients who are diagnosed with invasive ovarian epithelial adenocarcinoma or papillary serous fallopian tube carcinoma (no low malignant potential tumors) AND are without postoperative infection proceed to part B of the study.
* Part B: Patients undergo collection of postoperative serum specimen for proteomic profiling using SELDI/MALDI-TOF within 3-8 weeks after surgery, before starting chemotherapy, and at end of chemotherapy.

After completion of study procedures, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Abnormal pelvic mass by physical examination or imaging test

  * Undiagnosed
* Planning to undergo surgical evaluation within the next 3 weeks

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Proteomic proflie (i.e. discrimination of tumor from nontumor in pelvic mass)

CONTACTS AND LOCATIONS:
Overall Officials: Elise C. Kohn, MD, Study Chair — NCI - Medical Oncology Branch; Samir N. Khleif, MD — National Cancer Institute (NCI); Larry J. Copeland, MD — Ohio State University Comprehensive Cancer Center
Locations (107):
- United States (107):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Florida Gynecologic Oncology - Fort Myers, Fort Myers, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Chicago Gynecologic Oncology, Palatine, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Union Hospital Cancer Program at Union Hospital, Elkton Md, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center - Las Vegas, Las Vegas, Nevada
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Williamette Gynecologic Oncology PC, Portland, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Texas Medical Branch, Galveston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center at UV Health System, Charlottesville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Gynecologic Oncology Associates, Roanoke, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Aurora Women's Pavilion of West Allis Memorial Hospital, West Allis, Wisconsin